CLINICAL TRIAL: NCT00000525
Title: Diuretics, Hypertension, and Arrhythmias Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double
Other Study IDs: 44; R01HL036821 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Arrest; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Arrest; Heart Diseases; Hypertension | interventions — Hydrochlorothiazide; Diet; Triamterene; Chlorthalidone

INTERVENTIONS:
Drug: hydrochlorothiazide
Behavioral: diet, potassium supplementation
Behavioral: diet, magnesium supplementation
Drug: triamterene
Drug: chlorthalidone

SUMMARY:
To determine whether hypertensive patients with ECG abnormalities and receiving hydrochlorothiazide diuretics were at increased risk of sudden death.

DETAILED DESCRIPTION:
BACKGROUND:

The Multiple Risk Factor Intervention Trial (MRFIT) revealed an unexpected subgroup finding: an association between diuretic therapy (especially with hydrochlorothiazide) and an increased rate of sudden death in hypertensive men with left ventricular hypertrophy and other ECG abnormalities. The Diuretics, Hypertension, and Arrhythmias Clinical Trial sought to determine whether the finding resulted from random variation or represented a serious toxic response to hydrochlorothiazide.

DESIGN NARRATIVE:

Randomized, double-blind. Following one month of withdrawal from all diuretics and repletion with oral potassium and magnesium, the study participants were randomized to two months of treatment with one of six treatment groups: hydrochlorothiazide; hydrochlorothiazide with oral potassium; hydrochlorothiazide with oral potassium and magnesium; hydrochlorothiazide and triamterene; chlorthalidone; or placebo. The main outcome measures were ventricular arrhythmias on 24-hour Holter monitoring and serum and intracellular potassium and magnesium levels.

ELIGIBILITY:
Men, ages 35 to 70, with ECG abnormalities, diastolic blood pressure less than 95 mm Hg at entry.

Subjects had been treated for at least six months by their own physicians with hydrochlorothiazide (HCT), HCT and potassium supplementation, triamteren

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 1986-07; Primary Completion 1989-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hulley — University of California

REFERENCES:
- [Background] Siegel D, Cheitlin MD, Black DM, Seeley D, Hearst N, Hulley SB. Risk of ventricular arrhythmias in hypertensive men with left ventricular hypertrophy. Am J Cardiol. 1990 Mar 15;65(11):742-7. doi: 10.1016/0002-9149(90)91381-f. PMID 2138408
- [Background] Chang SW, Fine R, Siegel D, Chesney M, Black D, Hulley SB. The impact of diuretic therapy on reported sexual function. Arch Intern Med. 1991 Dec;151(12):2402-8. PMID 1746997
- [Background] Siegel D, Black DM, Seeley DG, Hulley SB. Circadian variation in ventricular arrhythmias in hypertensive men. Am J Cardiol. 1992 Feb 1;69(4):344-7. doi: 10.1016/0002-9149(92)90231-m. PMID 1734646
- [Background] Siegel D, Hulley SB, Black DM, Cheitlin MD, Sebastian A, Seeley DG, Hearst N, Fine R. Diuretics, serum and intracellular electrolyte levels, and ventricular arrhythmias in hypertensive men. JAMA. 1992 Feb 26;267(8):1083-9. PMID 1735925
- [Background] Siegel D, Cheitlin MD, Seeley DG, Black DM, Hulley SB. Silent myocardial ischemia in men with systemic hypertension and without clinical evidence of coronary artery disease. Am J Cardiol. 1992 Jul 1;70(1):86-90. doi: 10.1016/0002-9149(92)91395-k. PMID 1615875
- [Background] Siegel D, Saliba P, Haffner S. Glucose and insulin levels during diuretic therapy in hypertensive men. Hypertension. 1994 Jun;23(6 Pt 1):688-94. doi: 10.1161/01.hyp.23.6.688. PMID 8206564